CLINICAL TRIAL: NCT03577977
Title: Retrospective Data Collection on Betaferon Use in Children and Adolescents With Multiple Sclerosis
Brief Title: Betaferon Use in Children and Adolescents With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 2008/01743
Record Dates: First submitted 2018-06-25; First posted 2018-07-05 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis (MS), Betaseron, Betaferon
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with Betaferon: Patients with very early onset of MS, who received at least one injection of interferon beta-1b as prescribed by the treating physician, before the age of 18.
  Interventions: Drug: Interferon beta-1b (Betaseron, Betaferon, BAY86-5046)

INTERVENTIONS:
Drug: Interferon beta-1b (Betaseron, Betaferon, BAY86-5046) — Betaferon was injected subcutaneously as prescribed by the treating physician.

SUMMARY:
The objective of this study is to determine efficacy, safety and tolerability of interferon beta-1b for multiple sclerosis (MS) in children and adolescents

ELIGIBILITY:
Inclusion Criteria:

* patients with symptoms consistent with the diagnosis of a demyelinating CNS disease
* patients who received at least one injection of Betaferon before age 18 (before their 18th birthday)
* recorded use of at least one dose of Betaferon before January 1, 2008

Exclusion Criteria:

* Diagnosis other then MS or a demyelinating CNS disease

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Multiple sclerosis patients under 18 years old treated with at least one dose of Betaferon until 31.12.2007.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2008-06-01 (Actual); Primary Completion 2009-04-15 (Actual); Study Completion 2009-04-15 (Actual)

PRIMARY OUTCOMES:
Mean expanded disability status scale (EDSS) score at the end of trial participation | Up to 2 years
  The Expanded Disability Status Scale (EDSS) score is ranged between 1 (No disability, minimal signs in one Functional System) and 10 (death due to MS) measured in half-points on an ordinal scale.
Proportion of patients having the mean EDSS score of less than or equal to 3.0 and more than or equal to 3.5 at the end of the trial | Up to 2 years
  The Expanded Disability Status Scale (EDSS) score is ranged between 1 (No disability, minimal signs in one Functional System) and 10 (death due to MS) measured in half-points on an ordinal scale.
Mean frequency of complications recorded after start of betaferon therapy | Up to 2 years
Mean EDSS score on the exacerbations recorded after start of betaferon therapy | Up to 2 years
  The Expanded Disability Status Scale (EDSS) score is ranged between 1 (No disability, minimal signs in one Functional System) and 10 (death due to MS) measured in half-points on an ordinal scale.
Number of adverse events described during the trial and described as possibly, likely, or undoubtedly associated with the test drug | Up to 2 years
Number of mild, moderate, or severe adverse events | Up to 2 years
Number of serious adverse events described during the trial | Up to 2 years
Number of adverse events described during the trial and classified as an flu-like syndrome | Up to 2 years
Number of adverse events described during the trial and classified as a local reaction | Up to 2 years
Number of cases of betaferon discontinuation due to adverse events | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Russia